CLINICAL TRIAL: NCT05551065
Title: Prevalence of LVEF Non-recovery After Acute Myocardial Infarction
Brief Title: Post STEMI Echo Registry
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Gormin Tan gtan (Unknown)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Other Study IDs: 2022.038
Record Dates: First submitted 2022-09-16; First posted 2022-09-22 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST Elevation Myocardial Infarction; low Left Ventricular Ejection Fraction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Point-of-care ultrasound (POCUS) — Point-of-care ultrasound (POCUS) using a hand-held ultrasound (Vscan, GE Healthcare)

SUMMARY:
This is a prospective observational study of consecutive patients presenting with STEMI to the Prince of Wales Hospital over a 12-month period. All patients will receive standard of care including reperfusion and GDMT irrespective of study enrolment. Patient will be followed for 9 months after enrolled in this study. Point-of-care ultrasound (POCUS) using a hand-held ultrasound (Vscan, GE Healthcare) will be performed to assess baseline LVEF within 48 hours of admission. Patients with baseline moderate-to-severe LV dysfunction by visual POCUS assessment (i.e. LVEF <40%) will be recruited for follow-up LVEF assessment at 3 months. Patients with persistent LVEF <40% by POCUS will undergo formal echocardiography to confirm LVEF by either 2D area (Simpson's rule) and 3D volumetric measurements. In 9 month visit, patient's clinical data will be collected and no echo is needed during this visit.

DETAILED DESCRIPTION:
This is a prospective observational study of consecutive patients presenting with STEMI to the Prince of Wales Hospital over a 12-month period. All patients will receive standard of care including reperfusion and GDMT irrespective of study enrolment. Patient will be followed for 9 months after enrolled in this study. Point-of-care ultrasound (POCUS) using a hand-held ultrasound (Vscan, GE Healthcare) will be performed to assess baseline LVEF within 48 hours of admission. Patients with baseline moderate-to-severe LV dysfunction by visual POCUS assessment (i.e. LVEF <40%) will be recruited for follow-up LVEF assessment at 3 months. Patients with persistent LVEF <40% by POCUS will undergo formal echocardiography to confirm LVEF by either 2D area (Simpson's rule) and 3D volumetric measurements. In 9 month visit, patient's clinical data will be collected and no echo is needed during this visit.

Categorical variables were presented in frequency tables and were compared using the Pearson Chi square test if all cell sizes were more than 5, or Fisher exact test if otherwise. Parametric and nonparametric continuous variables were expressed as mean ± SD and median (interquartile range) and were compared using the Student t test and Mann-Whitney U test, respectively. P<0.05 was considered statistically significant. All statistical analyses were performed using SPSS version 24.0

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. STEMI (defined by symptoms of myocardial ischemia accompanied by persistent elevation of the ST segment on ECG and the subsequent rise of biomarkers of myocardial necrosis)
3. Ability to provide informed consent and to complete the study and required follow-up

Exclusion Criteria:

1. Pregnancy
2. Pre-existing ICD or CRT-D implantation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The medical records of patients who have STEMI will be reviewed to determine preliminary eligibility according to patient inclusion/exclusion criteria. After a patient signs an informed consent for this study, he/she is considered enrolled in the study. An informed consent including privacy authorization must be obtained prior to the enrollment. The signed Patient Informed Consent should be kept with the study documentation and must be available for monitoring.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-03 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) assessment | 9 months
  LVEF is equal or below 35% proved that patients have poor left ventricular ejection fraction.
  LVEF is 36-49% proved that ejection blood function of heart is below normal. LVEF is 50-75% proved that ejection blood function of heart is normal.

SECONDARY OUTCOMES:
Death | 9 months
  Death
NYHA heart failure class | 9 months
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  No NYHA class listed or unable to determine.
Valvular dysfunction | 9 months
  Valvular dysfunction defined as one or more of the valves in your heart doesn't work properly, as evident by echo results

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided